CLINICAL TRIAL: NCT02030860
Title: A Randomized Pilot/Pharmacodynamic/Genomic Study of Neoadjuvant Paricalcitol to Target the Microenvironment in Resectable Pancreatic Cancer
Brief Title: A Study of Neoadjuvant Paricalcitol to Target the Microenvironment in Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 23213
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Adenocarcinoma of the Pancreas
MeSH Terms: interventions — paricalcitol; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-operative Paricalcitol (Experimental): Subject will receive gemcitabine/abraxane with preoperatively paricalcitol. Patients randomized to receive paricalcitol pre-operatively will begin treatment with intravenous paricalcitol at 25 μg three times weekly for one cycle beginning day 1 of therapy until the day before surgery (+/- 3 days).
  Interventions: Drug: Paricalcitol; Drug: Abraxane; Drug: Gemcitabine
- No Pre-operative Paricalcitol (Active Comparator): Subject will receive gemcitabine/abraxane without paricalcitol preoperatively.
  Interventions: Drug: Abraxane; Drug: Gemcitabine

INTERVENTIONS:
Drug: Paricalcitol — Dose: 25 micrograms Route: IV Frequency (within a 28 day cycle):Three times weekly for one cycle beginning day 1 of therapy until the day before surgery (+/- 3 days) (for subjects randomized to receive paricalcitol), then three times weekly for 3 cycles post-operatively (for all subjects).
  Arms: Pre-operative Paricalcitol
Drug: Abraxane — Dose: 125mg/m2 Route: IV infusion over 30 minutes Frequency (within a 28 day cycle): Day 1, 8, 15
Drug: Gemcitabine — Dose: 1000mg/m2 Route: IV infusion over 30-100 minutes Frequency (within a 28 day cycle): Day 1, 8, 15

SUMMARY:
Study of neoadjuvant paricalcitol to target the microenvironment in resectable pancreatic cancer to determine the effect of targeting the vitamin D metabolic program in the tumors of patients treated with one cycle of gemcitabine/abraxane with or without paricalcitol prior to surgery for resectable pancreatic cancer.

DETAILED DESCRIPTION:
This study is a randomized pilot/pharmacodynamic/genomic study of neoadjuvant paricalcitol to target the microenvironment in resectable pancreatic cancer to determine the effect of targeting the vitamin D metabolic program in the tumors of patients treated with one cycle of gemcitabine/abraxane with or without paricalcitol prior to surgery for resectable pancreatic cancer through an assessment of cellular and imaging markers.

ELIGIBILITY:
Inclusion Criteria

* Previously untreated, apparently resectable, adenocarcinoma of the pancreas at registration.
* Age greater than or equal to 18 years
* Eastern Cooperative Oncology Group performance status of 0-2.
* Standard laboratory criteria for hematologic, biochemical, and urinary indices within a range that, in the opinion of the physician, clinically supports enrollment of the patient on the trial. Note: subjects must have: Creatinine < 2x Upper Normal Limit , Transaminases < 3x Upper Normal Limit, Neutrophils >1.5x109/L, and Platelets >100,000/mm3
* Ability to provide written informed consent

Exclusion Criteria

* Patients with hypercalcemia (blood levels greater than 11.5 mg/dL; in patients with kidney disease, blood calcium levels must be 9.5 mg/dL or lower before starting paricalcitol).
* Patients who are currently pregnant, planning to become pregnant, or breast-feeding.
* Patients who, in the opinion of the physician, would not be clinically appropriate for receipt of the therapy regimen associated with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years
  number of adverse events in 2years

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States